CLINICAL TRIAL: NCT01430052
Title: Randomized Phase II Study Comparing Gemcitabine/S-1 Combination Chemoradiotherapy With Gemcitabine/S-1 Combination Chemotherapy for Unresectable Locally Advanced Pancreatic Cancer.
Brief Title: Chemoradiotherapy With Gemcitabine/S-1 vs Gemcitabine/S-1 for Locally Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Osaka Medical Center for Cancer and Cardiovascular Diseases (Other)
Responsible Party: Principal Investigator, Tatsuya Ioka, Assistant director, Osaka Medical Center for Cancer and Cardiovascular Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TatsuyaIoka; UMIN000001990 (Registry Identifier: UMIN)
Record Dates: First submitted 2011-09-05; First posted 2011-09-07 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2015-04

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; S 1 (combination); titanium silicide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gemcitabine , S-1 (Other): Gemcitabine 1000mg/m2 on Day 1 and 8, every 3 weeks. S-1 60-100mg/day on Day 1 to 14, every 3 weeks
  Interventions: Drug: Drug: gemcitabine, S-1
- Gemcitabine, S-1, radiotherapy (Experimental): Gemcitabine 600mg/m2 on Day 1 and 8, every 3 weeks. S-1 60-100mg/day on Day 1 to 14, every 3 weeks with radiotherapy 50.4Gy in 28 fractions
  Interventions: Drug: gemcitabine, S-1, radiotherapy

INTERVENTIONS:
Drug: Drug: gemcitabine, S-1 — Gemcitabine 1,000mg/㎡ is administered with 30 min intravenous infusion on day 1 and 8 every 3 weeks. S-1 60mg/㎡/day is administered orally for 2 consecutive weeks every 3 weeks.
  Other Names: gemzer; TS-1
  Arms: Gemcitabine , S-1
Drug: gemcitabine, S-1, radiotherapy — Gemcitabine 600mg/㎡ is administered with 30 min intravenous infusion on day 1 and 8 every 3 weeks. S-1 60mg/㎡/day is administered orally for 2 consecutive weeks every 3 weeks. Concurrent radiotherapy (a total dose of 50.4Gy) was delivered in 28 fractions.
  Other Names: gemzer; TS-1
  Arms: Gemcitabine, S-1, radiotherapy

SUMMARY:
The purpose of this study is to evaluate the clinical effectiveness of Gemcitabine/S-1 combination chemoradiotherapy with Gemcitabine /S-1 combination chemotherapy for unresectable locally advanced pancreatic cancer.

DETAILED DESCRIPTION:
When cancer develops outside of the pancreas from within the anatomical placement of the pancreas itself, it becomes difficult to excise in most cases. Generally, most pancreatic cancers are already unresectable at the time of diagnosis when we have recognized infiltration of over 1/2 the circumference of major arteries such as the celiac artery and super mesenteric artery in particular.

In comparison with advanced pancreatic cancer with distant metastases, it is not easy to treat unresectable locally advanced pancreatic cancer, even when performing standard gemcitabine monotherapy. In the case of unresectable locally advanced pancreatic cancers without distant metastases, we are left with the choice of whether or not to perform radiation therapy. This decision remains unsolved worldwide, despite the continuing efforts of researchers to bring an end to the clinical doubt.

We will report our results as well as the problems of combining treatments with chemoradiotherapy, using the novel anticancer agent gemcitabine as well as/or S-1, not 5FU, predominantly from our own clinical trials on this occasion.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed adenocarcinoma, adenocarcinoma squamous carcinoma of pancreatic cancer.
2. Patients who confirmed unresectable locally advanced pancreatic cancer with the criteria below.

   * Involving over 1/2 circumference of major artery (SMA/CA). (Under 1/2 that was borderline lesion.)
   * Involving over the merging section of portal-SMV.
   * No distal metastasis with diagnostic imaging.
   * Confirmed by CT image performed with in four weeks before registration.
3. Performance Status:0-1(ECOG)
4. Patients of age =>20 and 80>
5. sufficient organ functions

   * neutrophils>=1,500/mm3
   * platelets>=100,000/mm3
   * hemoglobin>=9.0g/dl
   * AST(GOT)/ALT(GPT) <=150IU
   * total bilirubin <=2.0mg/dl, (or <=3.0mg/dl if biliary drainage were present)
   * serum creatinine <= 1.2mg/dl
   * creatinine clearance>=60ml/min
6. Life expectancy more than 3 months.
7. Written informed consent.

Exclusion Criteria:

1. Lung fibrosis or intestinal pneumonia, and anamnesis or imaging findings.
2. Watery diarrhea
3. Severe infection
4. Severe complication (heart failure, renal failure, hepatic insufficiency,hemorrhagic peptic ulcer, intestines paralysis,ileus or uncontrolled diabetes etc)
5. Massive pleural or abdominal effusion.
6. Metastasis to central nervous system.
7. Active synchronous or metachronous malignancy other than carcinoma in situ.
8. Regular use of flucytosine, fenitoin or warfarin
9. Pregnant or lactation women, or women with known or suspected pregnancy and men who want let to pregnancy
10. Severe mental illness
11. Patients who are judged inappropriate for the entry into the study by the investigator.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2009-04; Primary Completion 2012-12 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Two year survival rate | 2 years

SECONDARY OUTCOMES:
Progression free survival（PFS） | 4 years
Overall Survival (OS) | 4 years
Adverse events | 4 years
Response rate | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Tatsuya Ioka, MD, Study Director — Osaka Medical Center for Cancer and CVD
Locations (1):
- Osaka Medical Center for Cancer and Cardiovascular Diseases, Osaka, Japan